CLINICAL TRIAL: NCT00600509
Title: Bridging Study of L059(Levetiracetam) in Patients With Epilepsy by Double Blind Method
Brief Title: Bridging Study of L059 (Levetiracetam) in Patients With Epilepsy by Double Blind Method
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Collaborators: UCB Japan Co. Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N165
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Epilepsy
Keywords: Levetiracetam; Keppra
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levetiracetam

SUMMARY:
Double-blind, randomized, placebo-controlled, multi center trial to evaluate the efficacy and safety of levetiracetam as adjunctive treatment in adult Japanese epileptic subjects with partial onset seizures.

ELIGIBILITY:
Inclusion Criteria:

* simple and/or complex partial seizures with or without secondary generalization, and first partial seizure >= 2 years before selection visit;
* seizures classifiable according to the ILAE classification;
* minimum of 12 partial seizures per 12 weeks with a minimum of two partial seizures per 4 weeks from the selection visit to the end of the baseline period ;
* exposed to two or more standard AEDs;
* taking up to three of the standard AEDs, at the initiation of the trial.

Exclusion Criteria:

* medication influencing the CNS, except for medication taken for antiepileptic treatment;
* partial seizures uncountable due to clustering, including status epileptics, during the 3 months prior to the selection visit;
* history of cerebrovascular disease including transient ischemic attack (TIA) and progressive cerebral disorder or progressive neurological disorder;
* presence or history of any clinically significant allergic condition and complication or history of significant alcohol abuse or drug abuse in the past.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2001-01; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
partial onset seizure frequency per week | collection of seizure count throughout the whole study (baseline and treatment periods)

SECONDARY OUTCOMES:
safety and tolerability | safety and tolerability data were collected throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)